CLINICAL TRIAL: NCT01039454
Title: A Single-blind, Randomized, Placebo Controlled, Two-period Crossover fMRI Study to Investigate the Effects of the D3 Antagonist GSK598809 on Neural and Behavioural Responses to Food Reward and Reinforcement After a Single Oral Dose of GSK598809 in Overweight and Obese Subjects.
Brief Title: Effects of the D3 Antagonist GSK598809 on Food Reward and Reinforcement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 109710
Record Dates: First submitted 2009-12-10; First posted 2009-12-25 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Substance Dependence
Keywords: Food Reward; fMRI; Obese; Cognition; Food Addiction; Behaviour; Overweight; Food Reinforcement; Metabolic endpoints
MeSH Terms: conditions — Substance-Related Disorders; Obesity; Food Addiction; Behavior; Overweight | interventions — GSK598809

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 2 way cross over.
  Interventions: Drug: GSK598809 Placebo Capsules
- Active (Active Comparator): 2 Way cross over
  Interventions: Drug: GSK598809 Capsules

INTERVENTIONS:
Drug: GSK598809 Capsules — GSK598809 is being developed for the treatment of substance dependence and potentially other impulse control disorders.
  Arms: Active
Drug: GSK598809 Placebo Capsules — Treatment of substance dependence and potentially other impulse control disorders.
  Arms: Placebo

SUMMARY:
This novel compound is a new experimental treatment that may help people to stop compulsive overeating. Compulsive overeating or binge eating is one of the main reasons why people are overweight or obese. Recent research has shown that some kinds of overeating may be linked to a brain chemical called dopamine. There is some evidence that blocking the action of this chemical in animals can reduce food intake, particularly of foods that are high in fat and sugar. The purpose of this study is to find out if this compound (which blocks the effects of dopamine) has the same effect in overweight or obese people, as it does in animals.

DETAILED DESCRIPTION:
This novel compound is being developed for the treatment of substance dependence and potentially other impulse control disorders.

This is an fMRI study designed to examine the behavioural and physiological effects of a single dose of novel compound on food reward and reinforcement in relation to food seeking behaviour under conditions of fasting, using fMRI, neurocognitive and metabolic endpoints in overweight and obese subjects. These main objectives will be evaluated in the principal part of the study, Part A. The study will also consist of a follow up period of weight management with a dietician where exploratory objectives are considered, Part B.

Part A, will be a single-blind, randomised, placebo controlled, multi-centre, two-period cross-over study. Approximately 24 subjects will be enrolled such that a minimum of 20 subjects complete dosing and critical assessments. All subjects will be required to complete questionnaires, perform a series of behavioural tasks and scanning procedures. Safety and tolerability will be assessed by monitoring subjects for adverse events, vital signs, ECGs, movement disorders (EPS, Akathisia) and laboratory parameters. The pharmacokinetic profile of the compound in this subject population will be determined by blood sampling over a 72 hour period post dosing, in both sessions. Part B will consist of 12 weeks weight management directed by a dietician on an outpatient basis. Subjects will have fortnightly visits with a dietician and at the end of the 12 weeks complete three questionnaires (TFEQ-18R, DBEQ and YBOCS-BE) and have their weight measured to assess weight loss.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy
* right handed
* binge eating episode
* use appropriate contraception method
* willing to see a dietician
* overweight or obese (BMI 27 - 40 kg/m2)

Exclusion Criteria:

* pregnant or breast feeding female
* recent weight loss or gain
* recent use of weight loss drugs
* surgery for obesity
* abuse alcohol or drugs
* cannot do MRI scans
* smokers
* certain emotional problems being treated with medications
* medical, surgical or neuropsychiatric illness
* ECG abnormality
* sudden unexplained death or syncope in first degree relatives

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-12-18 (Actual); Primary Completion 2010-04-26 (Actual); Study Completion 2010-04-26 (Actual)

PRIMARY OUTCOMES:
Functional MRI: Food Processing Task, Food-Stop Signal Task, Food Stroop Task | 9 weeks
Behavioural Neurocognitive Task: Visual Probe Task, Stimulus Response Compatibility Task, Pavlovian-Instrumental Task. | 9 weeks

SECONDARY OUTCOMES:
Appetite VAS, Bond and Lader VAS, Distress VAS, BIS II, TFEQ, BIS/BAS, BDI-II, Body weight, Metabolic markers: plasma leptin, ghrelin, alpa MSH | 9 weeks
PK endpoints: AUC, Cmax, tmax, t1/2 | 9 weeks
Safety and tolerability: adverse events, laboratory values, cardiovascular - blood pressure; heart rate; ECGs, movement disorders, temperature, respiratory rate, serum prolactin, GH and TSH | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United Kingdom (2):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 109710 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/109710?search=study&search_terms=109710#rs
- Available data/document: Individual Participant Data Set: 109710 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109710 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109710 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109710 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109710 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109710 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register